CLINICAL TRIAL: NCT01882244
Title: Remotely Deployed Training for Cognitive Impairment Associated With TBI
Brief Title: Remotely Deployed TBI Study
Acronym: RD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RD2013-04-17
Record Dates: First submitted 2013-06-11; First posted 2013-06-20 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Brain Injury
Keywords: traumatic brain injury; cognition; rehabilitation; attentional regulation; working memory
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neural Pathfinder Training (Experimental): Neural Pathfinder training (PATH) will involve 6-8 weeks of training sessions with a trainer (1-2 hour sessions, average of 1 session per week), up to 3 hours of telephone contact with the trainer (about 15 minutes per week), and approximately 20 hours of home practice). Some subjects will only receive the PATH intervention.
  Interventions: Behavioral: Neural Pathfinder Training
- Brain Health Education (Active Comparator): Brain Health Education (EDU) will involve 6-8 weeks of training sessions with a trainer (1-2 hour sessions, average of 1 session per week), up to 3 hours of telephone contact with the trainer (about 15 minutes per week), and approximately 20 hours of home practice). Some subjects will only receive the EDU intervention. Some subjects will receive both the PATH and EDU interventions.
  Interventions: Behavioral: Brain Health Education

INTERVENTIONS:
Behavioral: Neural Pathfinder Training — Neural Pathfinder Training consists of game-based computerized training tools that target goal-directed attention regulation. Training will involve 6-8 weeks of 1-2 hour in-person or remote sessions with a trainer involving an average of one session per week; about 15 minutes a week of telephone contacts with the trainer; and approximately 20 hours of homework (35 minutes/5 days a week), consisting of short attentional regulation practice and computer-assisted cognitive training game play.
  Arms: Neural Pathfinder Training
Behavioral: Brain Health Education — Brain Health Education (EDU) will involve 6-8 weeks of 1-2 hour in-person or remote sessions covering brain anatomy and health with a trainer involving an average of one session per week; about 15 minutes a week of telephone contacts with the trainer; and approximately 20 hours of homework (35 minutes/5 days a week), consisting of computer game play involving decision-making and motor skills.
  Arms: Brain Health Education

SUMMARY:
Injury to the brain can change the core of a person's being, affecting brain functions necessary to accomplish important goals in a complex world. Deficits in attention, working memory, and other aspects of goal-directed cognition affect a broad range of pursuits in everyday life, and are among the most prevalent and long-lasting consequences of brain injuries. The objective of this research is to develop remotely deployed training tools that target the most common, persistent and debilitating cognitive functions affected by traumatic brain injury (TBI); test the potential effects of the intervention and compare these effects to an active comparison intervention; and determine the neurocognitive and functional effects of computer-assisted remote training.

DETAILED DESCRIPTION:
The objective of this research is to develop remotely deployed computer-assisted training interventions, including software tools and training protocols, to address cognitive neurologic impairment associated with TBI, improving cognitive functioning and thus increasing quality of life. These tools will be built on a strong foundation of cognitive neuroscience, empiric evidence and advanced clinical care, while addressing practical issues such as distance and therapist/patient time limitations. This research involves two phases: User testing and Assessment/Training.

Assessment and Training Assessments: The potential effects of remotely administered training will be assessed using neuropsychological tests of complex attention, executive function and memory, a test of functioning in challenging real world situations involving multitasking and goal management, and questionnaires assessing cognitive and emotional functioning in personal life.

Neurocognitive testing and functional evaluation sessions take 2- 3 hours each, or about 5 hours combined. The subject is free to take breaks throughout testing sessions, which will take place over one or two days. Subjects participate in assessments up to four times (Baseline, after 6-8 weeks; 12-16 weeks; and at 18-24 weeks), or up to 20 hours (5 hours x 4 time points). The investigators anticipate about 30 subjects will participate in assessments and training.

Experimental Intervention I: The Pathfinder training protocol will include supervised attentional regulation training sessions, either in-person or via the VA's video tele-health (VTEL) system, and home play of a computer game. Trainers will also call subjects between each supervised session to (i) check that patients are initiating home play (and help problem-solve or provide motivation, if necessary), and (ii) encourage transfer and generalization of learning, as per protocol. Home play will be configured to allow for about 35 minutes of play each day between supervised sessions. After the end of home game play, some additional time will be allowed for continued practice and application of trained skills in personal life.

Experimental Intervention II: Brain Health Education will consist of training sessions, either in-person or via the VA's video tele-health (VTEL) system, and home play of a computer game. The Brain Health Education protocol will be based on a curriculum already developed, designed to facilitate learning of TBI-relevant information. Trainers will also call subjects between each supervised session to (i) check that patients are initiating home play (and help problem-solve or provide motivation, if necessary). Home play will be configured to allow for about 35 minutes of play each day between supervised sessions. After the end of home game play, some additional time will be allowed for continued practice and review of TBI-relevant information.

Subjects will participate in either one or both experimental interventions, which are matched for time commitment. Participation in interventions will include weekly in-person or remote 1-2 hour sessions with a trainer over a period of 6-16 weeks. In addition to weekly training sessions, study activities will include about 15 minutes of weekly telephone contact with the trainer and about 35 minutes a day of playing a computerized game at home during the same period. Therefore, total training time range is approximately 43-93 hours, depending on whether participation includes one or both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a history of traumatic brain injury
* Age 24-65
* Mild residual dysfunction in executive control
* In the chronic, stable phase of recovery (>6 months from injury)
* On stable psychoactive medications (> 30 days)
* Able and willing to participate in training and assessments.

Exclusion Criteria:

* Unstable medical, neurologic or psychiatric conditions
* Severe cognitive dysfunction
* Ongoing illicit drug or alcohol abuse
* Severe depression, severe anxiety or severe PTSD precluding participation
* Poor English comprehension.

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2013-06; Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Goal Processing Scale Scores | Baseline, Week 6-8, Week 12-16, and Week 18-24
  Functional/Behavioral evaluation

SECONDARY OUTCOMES:
Change in Scores on Neuropsychological Assessment Measures | Baseline, Week 6-8, Week 12-16, and Week 18-24
  Battery of Neuropsychological Tests

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J-W Chen, MD, Principal Investigator — San Francisco VA Medical Center
Locations (2):
- United States (2):
  - VA Northern California Health Care System, Martinez, California
  - San Francisco VA Medical Center, San Francisco, California